CLINICAL TRIAL: NCT06663436
Title: A Phase 2 Single-Blind, Randomized, Controlled, Single Center Study to Assess the Immunogenicity and Safety of a 2-Dose Schedule With GVGH altsonflex1-2-3 Vaccine in African Infants (H06_02TP)
Brief Title: A Study on the Immune Response and Safety of a Multicomponent Shigella Vaccine in Preventing Shigellosis in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 219449
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diarrhoea
Keywords: Shigella; Shigellosis; altSonflex1-2-3; Infants; African; Safety; Immunogenicity
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary | interventions — Shigella Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Tetanus Toxoid; Hepatitis B Vaccines; Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- altSonflex1-2-3 Dose_A Group (Experimental): Participants randomized to receive altSonflex1-2-3 Dose A and MR-VAC on Day 1 and Day 169.
  Interventions: Biological: altSonflex1-2-3 Dose A; Biological: MR-VAC
- altSonflex1-2-3 Dose_B Group (Experimental): Participants randomized to receive altSonflex1-2-3 Dose B and MR-VAC on Day 1 and Day 169.
  Interventions: Biological: altSonflex1-2-3 Dose B; Biological: MR-VAC
- altSonflex1-2-3 Dose_C Group (Experimental): Participants randomized to receive altSonflex1-2-3 Dose C and MR-VAC on Day 1 and Day 169.
  Interventions: Biological: altSonflex1-2-3 Dose C; Biological: MR-VAC
- Control Group (Active Comparator): Participants randomized to receive TYPHIBEV on Day 1, Infanrix hexa on Day 169 and MR-VAC on Day 1 and Day 169.
  Interventions: Biological: TYPHIBEV; Combination Product: Infanrix hexa; Biological: MR-VAC

INTERVENTIONS:
Biological: altSonflex1-2-3 Dose A — altSonflex1-2-3 Dose A administered intramuscularly on Day 1 and Day 169
  Other Names: Shigella vaccine
  Arms: altSonflex1-2-3 Dose_A Group
Biological: altSonflex1-2-3 Dose B — altSonflex1-2-3 Dose B administered intramuscularly on Day 1 and Day 169
  Other Names: Shigella vaccine
  Arms: altSonflex1-2-3 Dose_B Group
Biological: altSonflex1-2-3 Dose C — altSonflex1-2-3 Dose C administered intramuscularly on Day 1 and Day 169
  Other Names: Shigella vaccine
  Arms: altSonflex1-2-3 Dose_C Group
Biological: TYPHIBEV — TYPHIBEV administered intramuscularly on Day 1
  Other Names: Biological E. Limited's Typhoid Vi-CRM197 conjugate vaccine
  Arms: Control Group
Combination Product: Infanrix hexa — Infanrix hexa administered intramuscularly on Day 169
  Other Names: GSK's Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated) and Haemophilus influenzae type b vaccine (adsorbed)
  Arms: Control Group
Biological: MR-VAC — MR-VAC co-administered subcutaneously on Day 1 and Day 169
  Other Names: Serum Institute of India's Measles and rubella vaccine (live)

SUMMARY:
This study evaluates the immune response and safety of a multicomponent, 2-dose Shigella vaccine in preventing shigellosis in African infants. The candidate vaccine, altSonflex1-2-3, is currently being evaluated in a Phase 2 age de-escalation (from least vulnerable adult population to most vulnerable paediatric population) clinical study in Kenya, with the aim of identifying a preferred dose, using a 3-dose vaccination schedule in infants from 9 months of age (NCT05073003). This Phase 2 clinical study will evaluate the safety and immunogenicity of an alternative 2-dose vaccination schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/ Legally acceptable representative (LAR), who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory assessment.
* Participants satisfying all screening requirements.
* Participants seronegative for hepatitis B, and hepatitis C.
* A male or female 9 months of age at the time of the first study intervention administration.
* Normal nutritional z-score.
* Previously completed routine childhood vaccinations to the best knowledge of the participant's parent(s)/LAR(s).
* Born at a gestation period of >=37 weeks to the best knowledge of the participant's parent(s)/LAR(s).
* Participants negative for human immunodeficiency virus as confirmed by DNA polymerase chain reaction testing.
* Participants negative for HLA-B27.

Exclusion Criteria:

* Known exposure to Shigella during lifetime of the participant as confirmed during interview with the participant's parent(s)/LAR(s) or documented by participant's records.
* Progressive, unstable, or uncontrolled clinical conditions.
* History (known or suspected) of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Major congenital defects, as assessed by the investigator.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity (known or suspected), including allergy, to medicinal products, vaccines, or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study.
* Acute disease and/or fever (defined as temperature >=38.0°C) at the time of enrollment.
* Any clinically significant hematological and/or biochemical laboratory abnormality.
* Confirmed positive COVID-19 test during the period starting 30 days before the first administration of study interventions (Day -30 to Day 1).
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) (Day -30 to Day 1), or their planned use during the study period.
* Planned administration/administration of a vaccine/product not foreseen by the Protocol in the period starting 21 days before the first dose and ending after the last dose of study intervention(s) administration with the exception of Coronavirus disease 2019 (COVID-19) vaccines and Expanded Program on Immunization (EPI) vaccines.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Prior receipt of an experimental Shigella vaccine or live Shigella challenge.
* Prior receipt of a Typhoid conjugate vaccine (TCV).
* Administration of immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, from birth or planned administration during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 days consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention drug or invasive medical device.
* Any study personnel or immediate dependents, family, or household member.
* Child in care.
* Participants who do not meet eligibility criteria for administration of control vaccines.

Ages: 39 Weeks to 43 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) of anti-serotype-specific Shigella lipopolysaccharides/O-antigen (LPS/OAg) serum Immunoglobulin G (IgG) | Day 1 (before administration of Dose 1)
GMTs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 169 (before administration of Dose 2)
GMTs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 29 (28 days after administration of Dose 1)
GMTs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 197 (28 days after administration of Dose 2)
Geometric mean concentrations (GMCs) of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 1 (before administration of Dose 1)
GMCs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 169 (before administration of Dose 2)
GMCs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 29 (28 days after administration of Dose 1)
GMCs of anti-serotype-specific Shigella LPS/OAg serum IgG | Day 197 (28 days after administration of Dose 2)
Number of infants with at least a 4-fold increase in anti-serotype-specific Shigella LPS/OAg serum IgG | Day 29 compared with baseline (Day 1)
Number of infants with at least a 4-fold increase in anti-serotype-specific Shigella LPS/OAg serum IgG | Day 197 compared with baseline (Day 1)
Number of infants with at least a 4-fold increase in anti-serotype-specific Shigella LPS/OAg serum IgG | Day 197 compared with pre-Dose 2 (Day 169)

SECONDARY OUTCOMES:
Number of infants with solicited administration-site events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 169)
  Solicited administration site events include pain, redness and swelling at administration site.
Number of infants with solicited systemic events | During 7 days after each study intervention administration (study interventions administered at Day 1 and Day 169)
  Solicited systemic events include fever. Fever is defined as temperature greater than or equal to (>=) 38.0°C and preferred location for measuring temperature is the axilla.
Number of infants with unsolicited adverse events (AEs) | During 28 days after each study intervention administration (study interventions administered at Day 1 and Day 169)
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of infants with serious adverse events (SAEs) during the entire study period | From Day 1 to Day 197
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongs existing hospitalization, results in disability/incapacity or other medically significant events.
Number of infants with deviations from laboratory reference values of hematological, renal, and hepatic panel test results | Day 8 compared with baseline (Day 1)
  Panel tests include measures of white blood cells, haemoglobin, platelets, neutrophils, creatinine, alanine aminotransferase (ALT), and aspartate aminotransferase (AST).
Number of infants with deviations from laboratory reference values of hematological, renal, and hepatic panel test results compared to pre-Dose 2 values | Day 176 compared with pre-Dose 2 (Day 169)
  Panel tests include measures of white blood cells, haemoglobin, platelets, neutrophils, creatinine, ALT, and AST.
Anti-measles IgG concentrations expressed as GMCs | At Day 1 (before the first MR-VAC vaccination) and Day 197 (28 days after the second MR-VAC vaccination)
Anti-rubella IgG concentrations expressed as GMCs | At Day 1 (before the first MR-VAC vaccination) and Day 197 (28 days after the second MR-VAC vaccination)
Number of infants with measles seroresponse >=150 mIU/mL and >=200 mIU/mL | At Day 197 (28 days after the second MR-VAC vaccination)
Number of infants with rubella seroresponse >=4 IU/mL and >=10 IU/mL | Day 197 (28 days after the second MR-VAC vaccination)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Kericho, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf